CLINICAL TRIAL: NCT03537781
Title: Nutritional Knowledge and the Effects of Hunger & Satiety on Snack Choice: a Randomised Controlled Trial
Brief Title: The Effect of Food Labelling and Satiety on Individuals Food Choice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Principal Investigator, Kim Wright, Research administrator, St Mary's University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMU_SHAS_2018_01.
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Food Preferences; Hunger
Keywords: food choice, food labels
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to a food labelling or no food labelling condition. Participants in each condition will be tested when hungry and when satiated
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food label available, hungry state (Experimental): foods will be displayed with food labels present and when participants had nothing to eat
  Interventions: Behavioral: Food labelling versus no food labelling
- food label available, satiated (Experimental): foods will be displayed with food labels present and when participants had already eaten breaksfast
  Interventions: Behavioral: Food labelling versus no food labelling
- food label unavailable, hungry state (Experimental): foods will be displayed without food labels present and when participants had nothing to eat
  Interventions: Behavioral: Food labelling versus no food labelling
- food label unavailable, satiated (Experimental): foods will be displayed without food labels present and when participants had already eaten breakfast
  Interventions: Behavioral: Food labelling versus no food labelling

INTERVENTIONS:
Behavioral: Food labelling versus no food labelling — Food labelling availability and satiety status

SUMMARY:
Previous research has shown that nutritional knowledge is a key indicator in healthy eating choices, but real-life examinations of the associations between both nutritional knowledge and state of hunger and satiety on individuals' food choice of healthy vs unhealthy snacks is limited.

The present study aims to investigate whether the presence of nutritional information on food labels will affect participants' food choice when hungry and when satiated.

DETAILED DESCRIPTION:
Previous research has shown that nutritional knowledge is a key indicator in healthy eating choices, but real-life examinations of the associations between both nutritional knowledge and state of hunger and satiety on individuals' food choice of healthy vs unhealthy snacks is limited.

As there is currently little research combining these facets, it would be interesting to investigate whether individuals who are provided with food labelling information would choose unhealthy snacks when hungry as than when satiated and whether this would differ for those who are not provided with food labelling information.

Based on this, the present study aims to investigate whether the presence of nutritional information in the form of food labels will affect participants' food choice when hungry and when satiated. The General Nutrition Knowledge Questionnaire will be used to assess participants baseline nutritional knowledge and will be used as a covariate in the research project.

ELIGIBILITY:
Inclusion Criteria: Male and females aged 18-65 years old; in general good health; not known allergies and any medical conditions (e.g. heart disease, asthma)

Exclusion Criteria: Those who are currently following a weight loss diet; have food allergies and any medical conditions which might restrict their food intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
food choice | 2 days
  participants will have to choose one snack from a choice of six differing on their fat content

CONTACTS AND LOCATIONS:
Overall Officials: Conor Gissane, PhD, Principal Investigator — St. Mary's University, Twickenham
Locations (1):
- St Marys University, London, United Kingdom